## **Borderline Personality Disorder and Emotion Regulation** Effects of emotion-focused vs. cognitive schema therapy interventions on emotion regulation deficits in borderline personality disorder - associations between clinical efficacy, brain network function and local glutamate/GABA metabolism Ethiks approval 04.06.2018, last time edited

Supplementary material - Information on assessment tools, reliability criteria and classification of Reliable Change Index (RCI) results

| Abbreviation | Inventory | Information | Reliability<br>(Cronbach's<br>alpha) | Test-retest reliability |
|---|---|---|---|---|
| PF-TK (s) | Patient Questionnaire Day-<br>Clinic Jena<br>( <u>Patientenfragebogen</u><br><u>Tagesklinik</u> ) | Standardized assessment of patient's case history, including psychiatric/psychotherapeutic history | | |
| SEFP<br>assessed<br>with STIP-<br>5.1 (c) | Levels of Personality Functioning Scale (LPFS) (Criterion A) (Skala zur Erfassung des Eunktionsniveaus der Persönlichkeit) assessed with the Semi-Structured Interview for Personality Functioning DSM-5 (STiP-5.1) | Measures the impairments in personality functioning (Criterion A); enabling a dimensional assessment of the general severity of personality pathology (English version: Levels of Personality Functioning Scale, LPFS) | α=.94 to .97<br>(Hutsebaut et al.,<br>2017) | not available<br>so far |
| PID-5 (s) | Personality Inventory for DSM-5 (Criterion B) (Persönlichkeits-Inventar für DSM-5) | Assessment of maladaptive personality traits | domain scales:<br>$\alpha$ =.84 to .96;<br>facets: $\alpha$ =.72 to<br>.96 (Al-Dajani et<br>al., 2015) | r <sub>tt</sub> = .92 to .95<br>(Dhillon &<br>Bagby, 2015) |
| BPDSI-IV (c) | Borderline Personality Disorder Severity Index (fourth edition) | DSM-IV based semi-structured interview that assesses frequency and severity of borderline manifestations during the last three months; interview is appropriate for repeated measurements and therefore for treatment evaluation. | α=.96 (Kröger et<br>al., 2013) | r <sub>tt</sub> =.72 to .77<br>(Arntz et al.<br>2003) |
| EHI (s) | Edinburgh Handedness Inventory | Most widely used handedness inventory | α=.95 (Veale,<br>2014) | |
| IDA-R | <u>Integrierte Diagnose der ADHS</u><br>im Erwachsenenalter | Well-established screening instrument for ADHD in adulthood | α=.86 (Retz et al.,<br>2013) | |
| WAIS-IV | <u>W</u> echsler <u>A</u> dult <u>I</u> ntelligence<br><u>S</u> cale (fourth version) | Well-established scale to assess cognitive ability in adults | α=.97 (Wechsler, 2008) | |
| CTQ (s) | <u>C</u> hildhood <u>T</u> rauma<br><u>Q</u> uestionnaire | Screening measure for history of childhood maltreatment | α=.94 (Wingenfeld et al., 2013) | |
| ERI (s) | Emotion Regulation Inventory (Emotionsregulations-Inventar) | Follows the Process Model of<br>Emotion Regulation proposed by<br>James Gross; primary outcome<br>measure | α=.82 (König,<br>2011) | $r_{tt}$ =.62 to<br>$r_{tt}$ =.80 (König, 2011) |
| FSVV (s) | Questionnaire concerning self-<br>harming behavior ( <u>F</u> ragebogen<br>zu <u>selbstverletzendem</u><br><u>V</u> erhalten) (modified version) | Gathers information about nature of self-harming behavior, triggers, consequences, indirect methods and destabilizing factors; <b>primary outcome measure</b> | not available so far | r <sub>tt</sub> =.63 to .84<br>(frequency)<br>(Reicherzer &<br>Brandl, 2011) |
| BSL-95 (s) | Borderline Symptom List ( <u>B</u> orderline- <u>S</u> ymptom- <u>L</u> iste) | Self-rating instrument for specific assessment of borderline-typical symptomatology; sensitivity for change according to therapy; secondary outcome measure (BPD-specific) | α=.97 (Bohus et<br>al., 2007) | r <sub>tt</sub> =.84 (Bohus<br>et al., 2007) |
| IIP-D (s) | Inventory of Interpersonal Problems ( <u>I</u> nventar zur Erfassung <u>i</u> nterpersonaler <u>P</u> robleme) | Measures distress arising from interpersonal sources; secondary outcome measure (BPD-specific) | α=.71 to .82<br>(Horowitz et al.,<br>2000) | r <sub>tt</sub> =.81 to .90<br>(Horowitz et<br>al., 2000) |
| FGG (s) | Questionnaire of thoughts and feelings ( <u>F</u> ragebogen zu <u>G</u> edanken und <u>G</u> efühlen) | Assessment of borderline-specific cognitions; based on cognitive models and Linehan's biosocial model of BPD; secondary outcome measure (BPD-specific) | α=.97 (Renneberg<br>& Seehausen,<br>2010) | r <sub>tt</sub> =.96 in BPD<br>(Renneberg &<br>Seehausen,<br>2010) |

| SMI (s) | Schema Mode Inventory (118 item version) ( <u>S</u> chema- <u>M</u> odus-<br>Inventar) | Measures the presence and intensity of the 14 schema modes; secondary outcome measure (BPD-specific) | α=.85 (Reiss et al.,<br>2011) | r <sub>tt</sub> =.84<br>(Lobbestael et<br>al., 2010) |
|---|---|---|---|---|
| YSQ-s3r (s) | Young Schema Questionnaire (third version, short form) | Measure of early maladapative schemas (that are theoretically and empirically linked with personality disorder features); secondary outcome measure (BPD-specific) | α=.70 to .91 for 17<br>of the 18 scales<br>(Kriston et al.,<br>2012) | r <sub>tt=</sub> .70 to .89 for<br>17 of the 18<br>schemas<br>(Phillips et al.,<br>2017) |
| BDI-II (s) | Beck Depression Inventory-II (Beck Depressionsinventar-II) | Assessing the intensity of depressive symptoms; items are congruent with the depression criteria of the DSM-IV | α= .84 to .90<br>(Kühner et al,<br>2007) | r <sub>tt</sub> = .78 (Kühner<br>et al, 2007) |
| SCL-90-R (s) | Symptom Checklist-90-Revised | Evaluation/Screening of <b>general psychopathology</b> within the past 7 days | α=.96 to .98<br>(Franke, 2002) | r <sub>tt</sub> = .69 to .92<br>(Franke, 2002) |
| FEP-2 (s) | Questionnaire to evaluation psychotherapeutic processes (Fragebogen zur Evaluation von Psychotherapieverläufen) | Monitoring of change and progress in psychotherapeutic and psychiatric interventions; measures 4 dimensions of therapeutic outcome | α=.74 to .94 (Lutz<br>et al., 2009) | r <sub>tt</sub> =.69 to .77<br>(Lutz et al.,<br>2009) |
| INEP (s) | Inventory for the Assessment of Negative Effects of Psychotherapy (Inventar zur Erfassung Negativer Effekte von Psychotherapie) | self-report instrument for assessing negative effects of psychotherapy | α=.86 (Ladwig et al, 2014) | |

Proposed terms to classify the Reliable Change Index and Clinical Significance (Wise, 2004)

| Reliable | Clinical Significance and Normative Change Criterion | | | |
|---|---|---|---|---|
| Change<br>Indexes | Confidence Levels (%) | Change of 2 SDs | Change of 1 SD | Change of 0.5 SD |
| 1.96 | 95 | Recovered | (+) Response | (+) Minimal Response |
| 1.28 | 90 | Remitted | (+) Response | (+) Minimal Response |
| 0.84 | 80 | Improved | (+) Partial Response | (+) Minimal Response |
| -0.84 | 80 | Mildly Deteriorated | (-) Partial Response | (-) Minimal Response |
| -1.28 | 90 | Moderately<br>Deteriorated | (-) Response | (-) Minimal Response |
| -1.96 | 95 | Deteriorated | (-) Response | (-) Minimal Response |